CLINICAL TRIAL: NCT05162859
Title: Exercise Training in Heart Failure With Preserved Ejection Fraction - a Long-term Follow-up
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 627/21 S
Record Dates: First submitted 2021-11-11; First posted 2021-12-17 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Former Exercise Training: Patients that were randomized to high-intensity-interval training, moderate continuous training (OptimEx-Clin) or moderate continuous training + resistance training (Ex-DHF)
- Former Control: Patients that were randomized to guideline control (OptimEx-Clin) or usual care (Ex-DHF)

SUMMARY:
Exercise training is an effective therapy for patients with heart failure with preserved ejection fraction. However, it is unclear, whether a one-year intervention has a sustainable effect beyond the active study phase. Hence, this study is a long-term follow-up of patients that were recruited for the OptimEx-Clin and Ex-DHF trials in Munich.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were previously randomized to OptimEx-Clin or Ex-DHF in Munich
* Written informed consent

Exclusion Criteria:

* Pregnancy / breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with heart failure with preserved ejection fraction that were included in previous exercise intervention trials in Munich, Germany (OptimEx-Clin, NCT02078947; Ex-DHF, ISRCTN86879094)
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (mL/kg/min) | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)

SECONDARY OUTCOMES:
Change in oxygen consumption at the first ventilatory threshold (mL/kg/min) | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)
Change in ventilation-to-carbon-dioxide production slope | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)
Change in E/e' | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)
Change in left ventricular ejection fraction (%) | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)
Change in quality of life | From Baseline Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 4.6 to 9.1 years)
  Changes in Short Form-36 questionnaire (patients from Ex-DHF, scale 0-100, higher is better) and Kansas City Cardiomyopathy Questionaire - Quality of Life domain (patients from OptimEx, scale 0-100, higher is better) will be combined using the standardized mean difference
Time to first cardiovascular event | From Last Visit of Ex-DHF / OptimEx to Long-Term Follow-Up (between 3.3 to 8.2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Fegers-Wustrow, MD, Principal Investigator — Klinikum rechts der Isar, Technical University of Munich; Stephan Mueller, Principal Investigator — Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Klinikum rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueller S, Winzer EB, Duvinage A, Gevaert AB, Edelmann F, Haller B, Pieske-Kraigher E, Beckers P, Bobenko A, Hommel J, Van de Heyning CM, Esefeld K, von Korn P, Christle JW, Haykowsky MJ, Linke A, Wisloff U, Adams V, Pieske B, van Craenenbroeck EM, Halle M; OptimEx-Clin Study Group. Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity Advice on Peak Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):542-551. doi: 10.1001/jama.2020.26812. PMID 33560320
- [Background] Suchy C, Massen L, Rognmo O, Van Craenenbroeck EM, Beckers P, Kraigher-Krainer E, Linke A, Adams V, Wisloff U, Pieske B, Halle M. Optimising exercise training in prevention and treatment of diastolic heart failure (OptimEx-CLIN): rationale and design of a prospective, randomised, controlled trial. Eur J Prev Cardiol. 2014 Nov;21(2 Suppl):18-25. doi: 10.1177/2047487314552764. PMID 25354950
- [Background] Edelmann F, Bobenko A, Gelbrich G, Hasenfuss G, Herrmann-Lingen C, Duvinage A, Schwarz S, Mende M, Prettin C, Trippel T, Lindhorst R, Morris D, Pieske-Kraigher E, Nolte K, Dungen HD, Wachter R, Halle M, Pieske B. Exercise training in Diastolic Heart Failure (Ex-DHF): rationale and design of a multicentre, prospective, randomized, controlled, parallel group trial. Eur J Heart Fail. 2017 Aug;19(8):1067-1074. doi: 10.1002/ejhf.862. Epub 2017 May 17. PMID 28516519